CLINICAL TRIAL: NCT02951572
Title: Non-invasive Ventilation and Physical Activity in Patients With Neuromuscular Disorders and Thoracic Wall Disorders
Brief Title: Non-invasive Ventilation and Physical Activity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problem
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Dries Testelmans, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S54220
Record Dates: First submitted 2013-12-09; First posted 2016-11-01 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Neuromuscular Diseases
Keywords: Noninvasive Ventilation; Physical activity
MeSH Terms: conditions — Neuromuscular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with RLD initiating NIV (Other): Patients with RLD initiating NIV according to Belgian Health guidelines are followed-up before and after NIV initiation
  Interventions: Device: NIV

INTERVENTIONS:
Device: NIV

SUMMARY:
As fatigue and daytime sleepiness are typical symptoms of alveolar hypoventilation in patients with neuromuscular disorders and thoracic deformations, we hope, by starting non-invasive ventilation and improving these symptoms, to increase their physical activity.

DETAILED DESCRIPTION:
Patients with neuromuscular disorders and thoracic deformations develop alveolar hypoventilation during their disease progression. At that time, non-invasive ventilation(NIV) can be started as treatment.

Fatigue and daytime sleepiness are typical symptoms of alveolar hypoventilation. NIV has the intention to improve these symptoms but no research has been performed whether these improvements also objectively improve physical activity. Further on, no research has been performed on muscle strength and muscle fatigue.

Patients' physical activity, physical capacity and sleep quality will be measured before NIV initiation, after 3 months and 1 year of NIV use.

To start NIV, patients will be admitted to our sleep laboratory for 5 days/4 nights. Polysomnography will be used during NIV titration.

Physical activity will each time be measured by 2 activity monitors during 5 days.

ELIGIBILITY:
Inclusion Criteria:

* restrictive pulmonary function test AND
* symptoms of nocturnal alveolar hypoventilation or
* increased daytime pressure of arterial CO2 (PaCO2) (>45 mmHg) or
* >= 10 mmHg increase in PaCO2 during sleep in comparison to a normal awake supine value

Exclusion Criteria:

* patients < 16 years
* severe cardiac arrythmias or conduction disturbances
* severe mental disturbances
* amyotrophic lateral sclerosis
* total wheelchair-dependent patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Average daily walking time | Measured before initiation of NIV
  Average daily walking time will be measured by the McRoberts physical activity monitor
Average daily walking time | Measured after 3 months of NIV
  Average daily walking time will be measured by the McRoberts physical activity monitor
Average daily walking time | Measured after 1 year of NIV
  Average daily walking time will be measured by the McRoberts physical activity monitor

SECONDARY OUTCOMES:
Change in functional exercise capacity | Before NIV initiation
  Six minute walking test
Change in muscle strength | Before NIV initiation
  Quadriceps muscle strength will be measured by magnetic stimulation. MicroFet measurements of wrist flexion/extension and ankle dorsiflexion/plantar flexion Respiratory muscle strength will be measured by maximal inspiratory pressure and sniff nasal inspiratory pressure
Change in quadriceps fatiguability | Before NIV intiation
  Use of magnetic stimulation before and after performing fatigue test of the quadriceps muscle
Change in sleep structure and quality of sleep | Before NIV intiation
  Full polysomnography will be used to get insight in sleep improvement
Change in functional exercise capacity | After 3 months of NIV use
  Six minute walking test
Change in functional exercise capacity | After 1 year NIV use
  Six minute walking test
Change in muscle strength | After 3 months of NIV use
  Quadriceps muscle strength will be measured by magnetic stimulation. MicroFet measurements of wrist flexion/extension and ankle dorsiflexion/plantar flexion Respiratory muscle strength will be measured by maximal inspiratory pressure and sniff nasal inspiratory pressure
Change in muscle strength | After 1 year NIV use
  Quadriceps muscle strength will be measured by magnetic stimulation. MicroFet measurements of wrist flexion/extension and ankle dorsiflexion/plantar flexion Respiratory muscle strength will be measured by maximal inspiratory pressure and sniff nasal inspiratory pressure
Change in quadriceps fatiguability | After 3 months of NIV use
  Use of magnetic stimulation before and after performing fatigue test of the quadriceps muscle
Change in quadriceps fatiguability | After 1 year NIV use
  Use of magnetic stimulation before and after performing fatigue test of the quadriceps muscle
Change in sleep structure and quality of sleep | After 3 months of NIV use
  Full polysomnography will be used to get insight in sleep improvement
Change in sleep structure and quality of sleep | After 1 year NIV use
  Full polysomnography will be used to get insight in sleep improvement

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Bertien Buyse, MD,PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium